CLINICAL TRIAL: NCT07078591
Title: Phase 2 Study of Venetoclax-containing Therapy in Combination With HLA-mismatched Mobilized Peripheral Blood Mononuclear Cell Infusion for Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Venetoclax-containing Therapy Combined With Microtransplant for Newly Diagnosed AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEN-MST for AML
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: venetoclax; microtransplant; microtransplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants fit for intensive therapy (Experimental): This cohort will include patients fit for intensive therapy.
  Induction phase:
  Genetically low-risk patients Venetoclax 100mg on Day 4, 200mg on Day 5, 400mg on Days 6-11 orally; Daunorubicin 60mg/m2 or idarubicin 12mg/m2 IV daily on Days 1-3; Cytarabine 100mg/m2 IV daily on Days 1-7. No more than two cycles. Continue to consolidation phase if achieving CR/CRi.
  Genetically intermediate/high-risk patients Venetoclax 100mg on Day 1, 200mg on Day 2, 400 mg on Days 3-28 orally; Azacitidine 75mg/m2 SC daily on Days 1-7. 28 days per cycle, and no more than two cycles. Continue to consolidation phase if achieving CR/CRi and refuse allogeneic HSCT.
  Consolidation phase:
  Patients < 60 years Cytarabine 1.5g/m2 IV every 12 hours on Days 1, 2, 3; Venetoclax 400mg on Days 1-7. Infuse donor GPBMCs on Day 8. Totally 3-4 cycles.
  Patients ≥ 60 years Cytarabine 1g/m2 IV every 12 hours on Days 1, 2, 3; Venetoclax 400mg on Days 1-7. Infuse donor GPBMCs on Day 8. Totally 3-4 cycles.
  Interventions: Drug: Venetoclax; Drug: Azacitidine (AZA); Drug: Daunorubicin; Drug: Idarubicin（IDA）; Drug: Cytarabine (Ara-C); Biological: GPBMC infusion
- Participants unfit for intensive therapy but fit for lower intensity therapy (Experimental): This cohort will include patients unfit for intensive therapy but fit for lower intensity therapy at diagnosis according to Ferrara 2013 criteria.
  Induction phase:
  Venetoclax 100mg on Day 1, 200mg on Day 2, 400 mg on Days 3-28 orally; Azacitidine 75mg/m2 SC daily on Days 1-7. 28 days per cycle, and no more than two cycles. Re-evaluate unfitness and continue to consolidation phase if achieving CR/CRi and refuse allogeneic HSCT.
  Consolidation phase:
  Convert to "fit" patients and < 60 years Cytarabine 1.5g/m2 IV every 12 hours on Days 1, 2, 3; Venetoclax 400mg on Days 1-7. Infuse donor GPBMCs on Day 8. Totally 3-4 cycles.
  Convert to "fit" patients and ≥ 60 years Cytarabine 1g/m2 IV every 12 hours on Days 1, 2, 3; Venetoclax 400mg on Days 1-7. Infuse donor GPBMCs on Day 8. Totally 3-4 cycles.
  Still "unfit" patients Venetoclax 400 mg on Days 1-14 orally; Azacitidine 75mg/m2 SC daily on Days 1-7. Infuse donor GPBMCs on Day 15. 28 days per cycle until progression or untolerated.
  Interventions: Drug: Venetoclax; Drug: Azacitidine (AZA); Drug: Cytarabine (Ara-C); Biological: GPBMC infusion

INTERVENTIONS:
Drug: Venetoclax — Given PO
Drug: Azacitidine (AZA) — Given SC
Drug: Daunorubicin — Given IV
  Arms: Participants fit for intensive therapy
Drug: Idarubicin（IDA） — Given IV
  Arms: Participants fit for intensive therapy
Drug: Cytarabine (Ara-C) — Given IV
Biological: GPBMC infusion — HLA-mismatched donor GPBMC infusion

SUMMARY:
The purpose of this study is to evaluate whether HLA-mismatched donor G-CSF mobilized peripheral blood mononuclear cell (GPBMC) infusion with venetoclax-containing regimens (microtransplant, MST) could improve survival in adult patients with newly diagnosed acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, male or female, non-limited by race or ethnicity.
* No prior anti-acute leukemia treatment (including hypomethylators for leukemia or MDS) with the exception that prior hydroxyurea and/or leukapheresis are permitted.
* Confirmed acute myeloid leukemia in accordance with WHO criteria with a WBC count < 25 × 109/L.
* Adequate hepatic function including alanine transaminase (ALT) and aspartate aminotransferase (AST )<= 3 × upper limit of normal(ULN), and total bilirubin <= 1.5 × ULN.
* Adequate renal function including serum creatinine <= 2 × ULN or CrCl>= 40mL/min.
* LVEF measured by echocardiogram is within the normal range (LVEF > 50%).
* The subject must have one donor who is >= 18 years old and HLA matched at 0-7/10 loci (i.e., at least 3 HLA loci must be mismatched). In addition, the donor voluntarily donates hematopoietic stem cells and signs the consent form.
* Each subject (or his/her legal representatives) must sign the Informed Consent Form (ICF), indicating that he/she understands the purpose and procedures of research, and is willing to participate in research.
* Donor inclusion criteria: The donor meets the institution's criteria for related peripheral blood hematopoietic stem cell donors. The donor must be able to tolerate the cell separation and collection process, and sign the Informed Consent Form.

Exclusion Criteria:

* Acute promyelocytic leukemia, myeloid sarcoma, chronic myeloid leukemia accelerated phase and blast crisis.
* Uncontrolled infection or hemorrhage.
* Cardiovascular disease with clinical significance, such as uncontrolled or highly symptomatic cardiac arrhythmias, congestive heart failure, or myocardial infarction within 6 months prior to screening, or New York Heart Association (NYHA) function class 3 (moderate) or class 4 (severe) heart disease.
* Uncontrolled autoimmune disease or requiring immunosuppression treatment.
* History of severe blood infusion reaction.
* Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception.
* Psychiatric disorder or cognitive impairment that in the researcher's judgment would make the subject not likely to adhere to the protocol requirements.
* Any major surgery within 4 weeks before enrollment.
* Life-threatening illness other than AML or uncontrolled intercurrent illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Measured up to 4 years after the last participant is enrolled
  OS is defined as the number of days from the date of initiation of treatment to the date of death.
Event-free Survival (EFS) | Measured up to 4 years after the last participant is enrolled
  EFS is defined as the number of days from initiation of treatment to the date of progressive disease, relapse from CR or CRi, treatment failure or death from any cause.

SECONDARY OUTCOMES:
Complete remission (CR) and complete remission with incomplete marrow recovery (CRi) | Measured up to 2 years after the last participant is enrolled
  CR is defined as absolute neutrophil count > 1 × 109/L, platelet count > 100 × 109/L, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophil count <= 1 × 109/L or platelet count <= 100 × 109/L.
Partial remission (PR) | Measured up to 2 years after the last participant is enrolled
  PR is defined as decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow, peripheral blood neutrophil count > 1 × 109/L, platelet count > 100 × 109/L, red cell transfusion independence.
Non-relapse Mortality (NRM) | Measured up to 4 years after the last participant is enrolled
  NRM is defined as the death without relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Cai, MD, Principal Investigator — Department of Hematology, the Fifth Medical Center of Chinese PLA General Hospital
Locations (1):
- Department of Hematology, the Fifth Medical Center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No